CLINICAL TRIAL: NCT00190632
Title: Long-Term Monitoring of Safety in Subjects Treated With Duloxetine for Stress Urinary Incontinence
Brief Title: To Evaluate the Safety in Patients Taking Duloxetine for Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2690; F1J-MC-SBAY
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
This is an on-going study to evaluate the long-term safety and maintenance of effect of duloxetine in patients suffering with stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

Have had symptoms of SUI for at least 3 months prior to study entry.

Have urine leakage most often associated with activity (such as coughing, sneezing, exercise).

Ambulatory and able to use a toilet independently and without difficulty.

-

Exclusion Criteria:

Subjects who participated or were discontinued from any previous studies investigating duloxetine.

Use of excluded medications within 14 days prior to study entry or at any time during the study.

Subjects who currently have or have had a history of urogenital cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2001-03; Study Completion 2006-04

PRIMARY OUTCOMES:
To generate long-term safety data for duloxetine in the treatment of women with stress urinary incontinence (SUI)

SECONDARY OUTCOMES:
To collect data to demonstrate the maintenance of effect of duloxetine as measured by the Patient Global Impression of Improvement (PGI-I) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Cleveland, Ohio, United States